CLINICAL TRIAL: NCT02989155
Title: Tranexamic Acid Use and Blood Loss in Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Nicoleta Stoicea, Research Scientist/ Adj. Assistant Professor, Ohio State University
Other Study IDs: 2015H0427
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Tranexamic Acid Use; Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the need for a blood transfusion during surgery and to evaluate the levels of certain proteins in the blood when given tranexamic acid.

DETAILED DESCRIPTION:
A review of the medical record between January 01 2013 to July 1st 2015 will be used to determine if the hypothesis that patients receiving tranexamic acid will have a lower need for blood transfusion and there are changes in the levels of the proteins essential for healthy oxygen transport throughout the body is correct. Tranexamic acid is a medication which may help wounds to stop bleeding more quickly. Participants are not expected to receive any direct benefits from participating in this study. Only a small risk of private patient medical information being exposed is anticipated. The results of this study will help surgeons and the medical community to better understand the uses of this type of drug and its possible role in benefiting hip replacement patients during and following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age and older
* Surgical patients who underwent primary total hip arthroplasty (THA)
* Surgical patients who underwent revision THA
* Preoperative hemoglobin values (N) 11 g/dl
* Normal international normalized ratio (INR), prothrombin time (PT), partial thromboplastin time (PTT) values

Exclusion Criteria:

* - Allergy to tranexamic acid
* Bilateral THA
* History of ischemic heart disease
* Severe chronic heart failure
* Hepatic dysfunction
* Chronic renal failure
* On hemodialysis
* Cerebral infarction
* History of seizure
* Bleeding disorder
* Anticoagulant or aspirin-like medication and long acting NSAID medication
* Short acting NSAID's were discontinued at least 24 hrs before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four surgeons providing total hip replacement services within the date range for data collection have formally agreed to include their patients in the study population, therefore identification of patients will occur through screening the surgery log of each surgeon performing these surgeries within the defined date range.
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
hemoglobin, hematocrit, and red blood cell transfusion rates | Peri-operative care
  Whether intraoperative dose of 2gr tranexamic acid (TXA) in patients having primary or revision THA would decrease the perioperative and post-operative reduction in hemoglobin, hematocrit, and red blood cell transfusion rates compared with those of a similar group of patients who did not receive TXA (control group).

SECONDARY OUTCOMES:
clinically-significant venous thromboembolism (VTE) and all-cause mortality | within 30 days of surgery
  frequency of clinically-significant venous thromboembolism (VTE) and all-cause mortality within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nicoleta Stoicea, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No